CLINICAL TRIAL: NCT01504776
Title: A Phase I Study of Panobinostat in Combination With Bortezomib in the Treatment of Relapsed and/or Refractory Mantle Cell Lymphoma
Brief Title: Phase I Study of Panobinostat + Bortezomib for Relapsed and/or Refractory Mantle Cell Lymphoma (MCL)
Acronym: BUS48T
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anand Jillella (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Anand Jillella, Chief, Hematology/Oncology, Augusta University
Organization: Augusta University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589BUS48T
Record Dates: First submitted 2011-08-08; First posted 2012-01-05 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2012-01

CONDITIONS: Mantle Cell Lymphoma
Keywords: MCL; Lymphoma; Panobinostat
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — Panobinostat; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label Drug Therapy (Experimental): Single arm
  Interventions: Drug: Panobinostat; Drug: Bortezomib

INTERVENTIONS:
Drug: Panobinostat — Dose escalation study of oral panobinostat administered Monday-Wednesday-Friday (MWF) weekly x 4 weeks, utilizing 3+3 dosing scheme (15, 20, 25 mg) in combination with a fixed dose of bortezomib 1.3 mg/m2 administered as a short intravenous (IV)infusion of 3-5 seconds every week x 4 weeks, representing one cycle. Each week, bortezomib will be administered IV prior to the oral dose of panobinostat
  Other Names: LBH589
Drug: Bortezomib

SUMMARY:
The purpose of this study is to determine the safety and clinical efficacy of the combination of panobinostat plus bortezomib.

DETAILED DESCRIPTION:
This is a phase I single arm, open label, multi-center (3 participating sites) dose escalation study of oral panobinostat administered Monday-Wednesday-Friday (MWF) weekly x 4 weeks, utilizing 3+3 dosing scheme (15, 20, 25 mg) in combination with a fixed dose of bortezomib 1.3 mg/m2 administered as a short intravenous (IV) infusion of 3-5 seconds every week x 4 weeks, representing one cycle. Each week, bortezomib will be administered IV prior to the oral dose of panobinostat. There will be sub-investigators participating in this study who will enroll at sub-sites.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years old
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Patients must have adequate hematology/chemistry lab values
* Echocardiogram (ECHO) must demonstrate Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Patients with previously diagnosed MCL based on standard criteria and with at least one and a maximum of 4 lines of therapy and currently requiring further treatment
* Prior therapy with autologous and allogeneic stem cell transplant is permissible. Patients who have undergone an allogeneic transplant should have no evidence of graft-versus-host disease (GVHD) and should not be on any immunosuppressive therapy. Autologous and allogeneic transplant will be counted as one prior therapy.
* Patients previously treated with bortezomib will be included in the study

Exclusion Criteria:

* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 (Panobinostat) treatment
* Peripheral neuropathy ≥ Common Toxicity Criteria for Adverse Effects (CTCAE) grade 2 on clinical examination within 14 days of randomization
* Impaired cardiac function or clinically significant cardiac diseases
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of LBH589
* Patients with diarrhea > CTCAE grade 2.
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
* Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Patients who have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (whichever is longer) and who have not recovered from side effects of those therapies.
* Patients who have received either immunotherapy within < 8 weeks; chemotherapy within < 4 weeks; or radiation therapy to > 30% of marrow-bearing bone within < 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies.
* Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not using an effective method of birth control. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential must have a negative serum pregnancy test within 24hrs of receiving the first dose of study medication.
* Male patients whose sexual partners are WOCBP not using effective birth control
* Patients with a prior malignancy within the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
* Patients with known positivity for human immunodeficiency virus (HIV) ) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.
* Allergic reaction to bortezomib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD) | 3 years
  To determine the DLTs and MTD of panobinostat given in combination with bortezomib.

SECONDARY OUTCOMES:
Observe the activity of the combination against Mantle Cell Lymphoma (MCL) in patients treated in this Phase I study. | 3 years
  Pre-treatment primary MCL cells derived from the bone marrow and/or peripheral blood of patients enrolled in this clinical trial will be isolated and treated ex vivo with panobinostat and/or bortezomib. IC50 values for each agent, as well as the combination indices values for the two agents will be determined and correlated with clinical response.
  Pre-treatment and 24 hour post-treatment primary MCL cells from patients who have circulating MCL cells in the peripheral blood will be isolated, as above.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Jillella, MD, Principal Investigator — Augusta University
Locations (1):
- Georgia Regents University, Augusta, Georgia, United States